CLINICAL TRIAL: NCT01971372
Title: Comparing Methods of NSAID Delivery for Postoperative Pain
Brief Title: Post-Operative Pain Management With NSAIDS
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3411
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Urogynecologic Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aim 1: To identify differences in pain perception and satisfaction with pain control in women undergoing urogynecologic surgery receiving nonsteroidal anti-inflammatory (NSAIDS) postoperatively by oral ibuprofen, intravenous ibuprofen, or intravenous ketorolac. Specific Aim 2: To compare the differences in narcotic usage and medication side effects.

DETAILED DESCRIPTION:
All patient will be informed that they may receive either ibuprofen or ketorolac and that the medication may be given (IV) or per os (PO). Patients were also informed that their pain may improve or worsen during the study, and that they could request additional pain medication (as a rescue medication) at any time.

After surgery, all patients will be placed initially on a patient controlled analgesia (PCA) of hydromorphone with standardized settings of allowing the patient to dispense 0.2 mg of medication every 6 minutes (lockout rate) and an hourly maximum of 2.0 mg/hour. A one-time nursing bolus of 0.4 mg will also be ordered. The PCA will be discontinued on the morning after surgery no later than 12:00 noon. The patient will then be started on PO pain medication, either hydrocodone/acetaminophen or oxycodone/acetaminophen.

Immediately after surgery, patients will then be assigned to one of three treatment arms with a computer-generated randomization schedule that is to be based on their order of enrollment. Patients were informed they could withdraw at any point. Three visual analog scores (VAS) will be obtained from the patient before noon on the first day after surgery. One scale to assess pain at rest, one scale to assess pain with ambulation, and one scale to assess satisfaction with pain control.

The medications will each be given every 8 hours in order to keep all medications on a similar doing regimen. This will allow the patients to receive a total of three doses of medication over 24 hours, regardless of which arm of the study they are randomized to.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Available for reliable follow up
* Able to complete study assessment
* Scheduled for surgery by FPMRS surgeon

Exclusion Criteria:

* Age <18 years
* Known renal impairment
* Congestive heart failure
* Dementia or inability to follow instructions
* Allergy to NSAIDS
* Allergy to hydromorphone
* History of gastrointestinal bleeding or ulceration
* Inflammatory bowel disease

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited and consented through an IRB-approved process. Women and minorities are included in the research protocol. We will not exclude potential subjects from participating in this or any study solely on the basis of ethnic origin or socioeconomic status. There are no children involved in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain scores | Within 24 hours after surgery
  Three visual analog scores (VAS) will be obtained from the patient before noon on the first day after surgery. One scale to assess pain at rest, one scale to assess pain with ambulation, and one scale to assess satisfaction with pain control.

CONTACTS AND LOCATIONS:
Overall Officials: Mikio Nihira, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States